CLINICAL TRIAL: NCT02672696
Title: Interest of Navigation for the Treatment of Pertrochanteric Fractures With the Gamma 3 Nail
Acronym: INOPEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital du Valais (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fluoromap Gamma 3 nail
Record Dates: First submitted 2016-01-21; First posted 2016-02-03 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Femoral Fractures; Fracture Fixation, Internal; Trochanteric Fractures
Keywords: Navigation; Gamma Nail
MeSH Terms: conditions — Femoral Fractures; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FluoroMap group (Experimental): Adult patients with a proximal femoral fracture eligible for intramedullary nailing with a Gamma 3 nail (Stryker Inc).
  In this group, the surgeon will use the FluoroMap 3D reconstruction system (Stryker Inc) with the standard fluoroscopy to help him place the cephalic screw in the femoral head.
  Interventions: Device: FluoroMap 3D
- Test group (No Intervention): Adult patients with a proximal femoral fracture eligible for intramedullary nailing with a Gamma 3 nail (Stryker Inc).
  In this group, the surgeon will use only the standard fluoroscopy to help him visualize the position of the cephalic screw in the femoral head.

INTERVENTIONS:
Device: FluoroMap 3D — Use of the 3D reconstruction software developed by the manufacturer of the Gamma Nail (e.g. Stryker Inc.) along with the standard fluoroscopy
  Other Names: ADAPT System
  Arms: FluoroMap group

SUMMARY:
The aim of the study is to compare Tip-Apex Distance values in two groups of patients after intramedullary nailing of proximal femur. The first group of patients is operated with the help of a 3D reconstruction device connected to the standard fluoroscopy allowing the surgeon to visualize directly the exact position of the tip of the trans-cervical screw while the second group (which is the reference-group) is operated with the help of fluoroscopy alone.

DETAILED DESCRIPTION:
The main orthopedic complication after fixation of a proximal femoral fracture with a cephalo-medullary nail is the cut-out of the cephalic screw from femoral head resulting in a protrusion of this screw in the coxo-femoral joint, mostly during the first 6 months after the operation. In most cases, the surgeon has to remove the primary implant and perform a total hip arthroplasty to his patient, therefore rising the morbidity and social costs linked to the treatment of the initial fracture.

Baumgartner showed the importance of the position of the cephalic screw for predicting failure of the implant and proposed a new measurement to evaluate this position, the tip-apex distance which is the sum of the distance from the tip of the cephalic screw to the apex of the femoral head on an anteroposterior radiograph and this distance on a lateral radiograph, after controlling for magnification. He showed a lower TAD was associated with a lower risk of cut-out.

The aim of this study is to evaluate the help of a 3D reconstruction software linked to the standard fluoroscopy in achieving the lowest TAD and therefore minimizing the cut-out rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a proximal femoral fracture eligible for intramedullary nailing with a Gamma 3 Nail

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Tip-Apex distance | 6 months
  Change of the value of the tip-apex distance at each follow-up control (6 weeks, 3 and 6 months) compared to the post-op value

SECONDARY OUTCOMES:
Cut-out of the cephalic screw | 6 months
  Visualization of a migration of the tip of the cervical screw outside the femoral head on one radiological incidence will be considered as a "cut-out" and reported in the final results

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital du Valais, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: No